CLINICAL TRIAL: NCT02137473
Title: Optimizing Mothers' Milk for Preterm Infants (OptiMoM) Program of Research: Study 2-Bovine vs. Human Milk-Based Fortifier Study
Brief Title: Bovine vs. Human Milk-Based Fortifier Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, Research Institute, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000044263
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Very Low Birth Weight Infant (<1250g)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bovine protein-based fortifier (Active Comparator)
  Interventions: Other: Bovine protein-based fortifier
- Human milk-based fortifier (Experimental)
  Interventions: Other: Human milk-based fortifier

INTERVENTIONS:
Other: Human milk-based fortifier
  Arms: Human milk-based fortifier
Other: Bovine protein-based fortifier
  Arms: Bovine protein-based fortifier

SUMMARY:
Most very low birth weight infants accumulate a nutrient deficit in hospital due to minimal nutrient reserves and elevated nutritional requirements which may contribute to poor outcome. Adding nutrients to human milk improves their nutritional status and growth, but it is unclear if adding bovine protein-based fortifiers as is the current standard of care has some unintended negative consequences to neonates. Infants will be randomized to have their feeds (mother's own milk or pasteurized donor breastmilk) nutrient enriched with a human milk-based fortifier or a bovine protein-based fortifier and will be followed in hospital to assess feeding tolerance, growth, gut inflammation, mother's milk and infant gut microbiome, and neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* <1250g birth weight
* Parent(s) or guardian(s) agree to use donor breastmilk if own mother's milk supply is insufficient

Exclusion Criteria:

* Infant receives formula or a nutrient fortifier prior to randomization
* >day 14 at the time of enrollment and enteral feeds have not commenced
* Infants with major congenital or chromosomal anomalies that could impact growth
* Enrollment in another research study affecting nutritional management during the feeding intervention
* Reasonable potential that the infant will be transferred to a neonatal intensive care unit where the study protocol will not be continued

Max Age: 2 Weeks | Sex: All
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Feeding tolerance | 84 days of age, hospital discharge or when able to consume two oral feeds a day without supplementation (e.g. tube feeding), whichever comes first
  Percentage of infants with a significant feeding interruption as defined by days feedings held for ≥12 hours OR feeds reduced by >50% (ml/kg/d) not due to a clinical procedure or transitioning to the breast

SECONDARY OUTCOMES:
Growth | 84 days of age, hospital discharge or when able to consume two oral feeds a day without supplementation (e.g. tube feeding), whichever comes first
  Daily weight measurements, weekly length measurements, weekly head circumference measurements, z-scores for anthropometric measures

OTHER OUTCOMES:
Other measures of feeding tolerance | 84 days of age, hospital discharge or when able to consume two oral feeds a day without supplementation (e.g. tube feeding), whichever comes first
  Percent and number of days of emesis, gastric aspirates >50% pre-feed volume, abdominal distension (>2 cm), percentage of infants where enteral feeding was terminated and parenteral nutrition had to be commenced, some assessment of the interruption of feeds, how long it takes to reach full enteral feeds (150 ml/kg/d)
Gut inflammation | 84 days of age, hospital discharge or when able to consume two oral feeds a day without supplementation (e.g. tube feeding), whichever comes first
Morbidity/mortality composite | 84 days of age, hospital discharge or when able to consume two oral feeds a day without supplementation (e.g. tube feeding), whichever comes first
  Necrotizing enterocolitis, late onset sepsis, chronic lung disease, severe retinopathy of prematurity, death
Bayley Scales of Infant and Toddler Development (BSID)-III | 18-24 months corrected age
  Cognitive, language and motor development as assessed by the BSID-III
Gut microbiota | 56 days of age or hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD RD, Principal Investigator — The Hospital for Sick Children, University of Toronto; Sharon L Unger, MD FRCPC, Principal Investigator — Mount Sinai Hospital, University of Toronto
Locations (18):
- Canada (18):
  - Izaak Walton Killam Health Centre, Halifax, Nova Scotia
  - William Osler Health System-Brampton, Brampton, Ontario
  - William Osler Health System-Etobicoke, Etobicoke, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Rouge Valley Health System, Toronto, Ontario
  - The Scarborough Hospital-General, Toronto, Ontario
  - The Scarborough Hospital-Birchmount, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - St Joseph's Health Centre, Toronto, Ontario

REFERENCES:
- [Derived] Asbury MR, Shama S, Sa JY, Bando N, Butcher J, Comelli EM, Copeland JK, Forte V, Kiss A, Sherman PM, Stintzi A, Taibi A, Tomlinson C, Unger S, Wang PW, O'Connor DL; OptiMoM Feeding Group. Human milk nutrient fortifiers alter the developing gastrointestinal microbiota of very-low-birth-weight infants. Cell Host Microbe. 2022 Sep 14;30(9):1328-1339.e5. doi: 10.1016/j.chom.2022.07.011. Epub 2022 Aug 19. PMID 35987195
- [Derived] Hopperton KE, Pitino MA, Walton K, Kiss A, Unger SL, O'Connor DL, Bazinet RP. Docosahexaenoic acid and arachidonic acid levels are correlated in human milk: Implications for new European infant formula regulations. Lipids. 2022 May;57(3):197-202. doi: 10.1002/lipd.12338. Epub 2022 Feb 15. PMID 35170053
- [Derived] Hopperton KE, Pitino MA, Chouinard-Watkins R, Shama S, Sammut N, Bando N, Williams BA, Walton K, Kiss A, Unger SL, Bazinet RP, O'Connor DL. Determinants of fatty acid content and composition of human milk fed to infants born weighing <1250 g. Am J Clin Nutr. 2021 Oct 4;114(4):1523-1534. doi: 10.1093/ajcn/nqab222. PMID 34254983
- [Derived] Hopperton KE, O'Connor DL, Bando N, Conway AM, Ng DVY, Kiss A, Jackson J, Ly L; OptiMoM Feeding Group; Unger SL. Nutrient Enrichment of Human Milk with Human and Bovine Milk-Based Fortifiers for Infants Born <1250 g: 18-Month Neurodevelopment Follow-Up of a Randomized Clinical Trial. Curr Dev Nutr. 2019 Nov 12;3(12):nzz129. doi: 10.1093/cdn/nzz129. eCollection 2019 Dec. PMID 32154499
- [Derived] O'Connor DL, Kiss A, Tomlinson C, Bando N, Bayliss A, Campbell DM, Daneman A, Francis J, Kotsopoulos K, Shah PS, Vaz S, Williams B, Unger S; OptiMoM Feeding Group. Nutrient enrichment of human milk with human and bovine milk-based fortifiers for infants born weighing <1250 g: a randomized clinical trial. Am J Clin Nutr. 2018 Jul 1;108(1):108-116. doi: 10.1093/ajcn/nqy067. PMID 29878061